CLINICAL TRIAL: NCT03777930
Title: Prospective Clinical Study of the Effect of Thalidomide Combined With Megestrol Acetate on Lymphocyte, Inflammatory Factor Regulation and Nutritional Status in Patients With Advanced Malignant Tumors
Brief Title: The Evaluation of Curative Effect on Treatment of Tumor Above Thalidomide Combined With Megestrol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Fifth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: shenzhenfifth 201807
Record Dates: First submitted 2018-08-25; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cancer, Therapy-Related
Keywords: thalidomide; megestrol acetate; tumor; lymphocyte; inflammatory cytokines; nutritional
MeSH Terms: conditions — Neoplasms, Second Primary; Neoplasms | interventions — Antineoplastic Agents; Thalidomide; Megestrol Acetate

STUDY DESIGN:
Intervention Model Description: 200 patients with advanced tumors with a predicted survival period of ≥2 months were selected, including 100 patients with chemotherapy indications (50 patients were divided into chemotherapy group and 50 patients were divided into chemotherapy combined with TH and MG group according to the random principle) and 100 patients without chemotherapy indications (50 patients were randomly divided into the best supportive treatment group and 50 patients were randomly divided into the best supportive treatment group with TH and MG according to the random principle). The chemotherapy alone group and the best supportive treatment group were the control group. The thalidomide and megestrol acetate administration groups were administered with thalidomide 100 mg qn po and megestrol acetate 0.16 qd po for 8 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- chemotherapy group (Experimental): the patients were recepted chemotherapy alone
  Interventions: Drug: Chemotherapy drugs
- chemotherapy combined with TH and MG group (Experimental): the patients were recepted chemotherapy combined with thalidomide and megestrol
  Interventions: Drug: thalidomide and megestrol acetate
- the best supportive treatment group (Experimental): the patients were recepted the best supportive without chemotherapy
  Interventions: Other: optimal support treatment
- the best supportive treatment combined with TH and MG group (Experimental): the patients were recepted the best supportive combined with thalidomide and megestrol without chemotherapy
  Interventions: Drug: thalidomide and megestrol acetate

INTERVENTIONS:
Drug: Chemotherapy drugs — According to the NCCN Guidelines
  Arms: chemotherapy group
Drug: thalidomide and megestrol acetate — The thalidomide and megestrol acetate administration groups were administered with thalidomide 100 mg qn po and megestrol acetate 0.16 qd po for 8 weeks
  Other Names: Chemotherapy drugs
  Arms: chemotherapy combined with TH and MG group
Other: optimal support treatment — Patients who cannot tolerate chemotherapy and other cancer treatments receive optimal support for 8 weeks
  Arms: the best supportive treatment group
Drug: thalidomide and megestrol acetate — The thalidomide and megestrol acetate administration groups were administered with thalidomide 100 mg qn po and megestrol acetate 0.16 qd po for 8 weeks
  Other Names: optimal support treatment
  Arms: the best supportive treatment combined with TH and MG group

SUMMARY:
To observe the effect of thalidomide combined with megestrol acetate on lymphocyte, inflammatory factor regulation and nutritional status in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
This study was to select 200 patients with advanced tumors with an estimated survival of ≥ 2 months. 50 patients were randomly assigned to each group. The patients were divided into chemotherapy group, chemotherapy combined with thalidomide and megestrol acetate group, The best supportive treatment group, the best supportive treatment combined with thalidomide and megestrol acetate group. The chemotherapy group and the best supportive treatment group were the control group. The combined group was administered continuously for 8 weeks according to thalidomide 100 mg qn po and megestrol acetate 0.16 qd po. Calculating the sum of the longest diameters of the target lesions from each patient before and 8 week after treatment. Patients in each group before treatment, 4th week, and 7th week were observed T cell subsets, B cell subsets, NK cell subsets and the expression of inflammatory cytokines. Through nutritional assessment Table (PG-SGA), Multidimensional Deficit Power Meter (MFSI-SF), Quality of Life Assessment Scale (EORTC QLQ-C30), Prognostic Assessment Form (GPS), Physical Status Assessment Form (ECOG) and lean body mass, upper arm muscle circumference and upper arm muscle area analysis of the effect of thalidomide combined with megestrol acetate on the nutritional status of patients with advanced cancer which reveal that thalidomide combined with megestrol acetate may improve the immune regulation and nutritional status of patients with advanced malignant tumors mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignant tumor confirmed by histopathology or cytology (hepatocarcinoma can be clinical diagnosis)
* Must be able to swallow pills
* The age of the tester ≥ 18 years old
* Gender is not limited
* Kamofsky score > 20 points
* Estimated survival period ≥ 2 months
* Childbearing age Women need negative pregnancy test
* Patients voluntarily sign informed consent and receive follow-up
* The tester can cooperate to observe adverse events and efficacy
* All of the above conditions can be included

Exclusion Criteria:

* Active upper digestive tract ulcers, obvious vomiting, chronic diarrhea, intestinal obstruction, malabsorption, etc; other patients have been known to affect drug absorption, distribution, metabolism or clearance
* 2 or more important organ dysfunction
* Thrombosis Embolism history, except for thrombosis caused by PICC
* Patients suspected of having a history of allergy to thalidomide tablets
* Any significant clinical and laboratory abnormalities that researchers believe affect safety evaluators, such as: uncontrollable activity Microbial infection, grade II or above peripheral neuropathy (NCI CTC AE v4.0), congestive heart failure, myocardial infarction within 6 months, chronic kidney disease, thyroid dysfunction etc, and acceptance may bring significant metabolic or weight changes Patients with clinical disposition
* Patients with mental disorders, affecting the efficacy of the assessor
* During the trial period and within 3 months after the end of the trial, the subject and his partner are not willing to contraception
* Any of the above can not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-10 (Estimated); Primary Completion 2020-10-10 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Imaging efficacy evaluation | before and 8 week after treatment
  Clinical response Based on the Response Evaluation Criteria Solid Tumors (RECIST), the therapeutic effect was divided into complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD). Investigators calculate the sum of the longest diameter of the target lesions from each patient by CT or MRI.

SECONDARY OUTCOMES:
Observing the expression of lymphocyte subsets | before , the fourth and the seventh weeks of treatment
  Patients were detected Lymphocyte subgroups of 2 ml peripheral blood by Flow cytometer (BD FACSCalibur), which inclunde the T cell subsets, NK cell subset, B cell subset(percentage)
Observing the expression of inflammatory factors | before , the fourth and the seventh weeks of treatment
  2 ml of peripheral blood was taken from each patient. Flow cytometry was used to detect changes of inflammatory factor expression which include the IL-2, IL- 4, IL-5, IL-6, IL-9, IL-10, IL-13, IL-17A, IL-17F, IL-21, IL-22, IFN-γ and TNF-α(ug/ml)
Nutritional assessment | before , the fourth and the seventh weeks of treatment
  Scored Patient-Generated Subjiective Global Assessment（PG-SGA）form was used in the present study. The total score of PG-SGA is summed by the following four subscale scores（A+B+C+D）. The first measurement score（A）is self-assessed by the subject and consists of the following four parts: Weight Table（0-4），Eating Situation Table（0-6），Symptom Table （0-22），Activity and Body Function Table（0-3）. The remaining three measurements are completed by trained registered clinical physicians， dieticians，and nurses: Scale of relationship between disease and nutritional needs（B）（0-6），Metabolic demand scale（C）（0-9），Physical examination scale（D）（0-24）. The scoring was controlled by one researcher (H.R). The lower scores represent a better outcome and the higher scores represent a worse outcome.

OTHER OUTCOMES:
Multidimensional deficient power assessment | before , the fourth and the seventh weeks of treatment
  Multidimensional deficient power assessment (MFSI-SF) was used in the present study. The MFSI-SF scale contains 30 subjects' subjective feelings，such as muscle soreness and memory loss. Subjects were scored according to the degree of each sensation (0-4). The MFSI-SF scale total score is the sum of each sensation score (0-120). The lower scores represent a better outcome and the higher scores represent a worse outcome.
Quality of life assessment | before , the fourth and the seventh weeks of treatment
  Quality of Life Assessment Table (EORTC QLQ-C30) was used in the present study. The Quality of Life Assessment Table contains 28 subjects' subjective feelings and symptoms，such as tiredness and diarrhea within one week (A)，and two other indicators: health status，quality of life within one week (B). Subjects were scored according to the degree of each sensation (A 0-4) and (B 1-7). The Quality of Life Assessment Table is divided into two parts: the first part of the total score (0-112); the second part of the total scores (2-14). In the first part of the total scores: the lower scores represent a better outcome and the higher scores represent a worse outcome. In the second part of the total scores: the higher scores represent a better outcome and the lower scores represent a worse outcome.
Prognostic assessment | before , the fourth and the seventh weeks of treatment
  The prognostic assessment by GPS scores which were calculated by detecting peripheral blood CRP and albumin from each tumor patients.
  GPS scores：CRP < 10 mg/l，albumin> 35g/l，GPS 0；CRP > 10 mg/l，albumin > 35 g/l，GPS 1；CRP > 10 mg/l，albumin < 35 g/l，GPS 2. The lower scores represent a better outcome and the higher scores represent a worse outcome.
Performance status assessment | before , the fourth and the seventh weeks of treatment
  The performance status of patients with cancer is measured by the clinician through the ECOG score form (score:0-5)
Lean body mass | before , the fourth and the seventh weeks of treatment
  Patient's waist circumference and weight were measured by trained registered clinical dietitians, and the measuring was controlled by one researcher (H.R). The researcher calculate lean body mass by measurements of waist circumference and body weight
Upper arm muscle circumference and upper arm muscle area | before , the fourth and the seventh weeks of treatment
  Patient's upper arm circumference and triceps skinfold thickness were measured by trained registered clinical dietitians, and the measuring was controlled by one researcher (H.R). The researcher calculate Upper arm muscle circumference and upper arm muscle area by measurements of upper arm circumference and triceps skinfold thickness

IPD SHARING:
Plan to Share IPD: No